CLINICAL TRIAL: NCT07123935
Title: Assessing the Safety & Efficacy of RenalGuard® Therapy in the Prevention of Cardiac Surgery Associated Acute Kidney Injury (CSA-AKI) - SAFEGUARD Study
Brief Title: Safety & Efficacy of RenalGuard® Therapy in the Prevention of Cardiac Surgery Associated Acute Kidney Injury
Acronym: SAFEGUARD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CardioRenal Systems, Inc. (Industry)
Collaborators: University Malaysia Medical Centre (Unknown); Institut Jantung Negara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RG-CSA-AKI-Malaysia-003
Record Dates: First submitted 2025-07-29; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Cardiac Surgery Associated - Acute Kidney Injury; AKI - Acute Kidney Injury
Keywords: acute kidney injury; cardiac surgery; RenalGuard Therapy; matched enhanced diuresis
MeSH Terms: conditions — Acute Kidney Injury | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Current Standard of Care
  Interventions: Other: Standard of Care (SOC)
- Study Group (Active Comparator): Patient with RenalGuard® Therapy
  Interventions: Device: RenalGuard® Therapy

INTERVENTIONS:
Device: RenalGuard® Therapy — RenalGuard Therapy®
  Arms: Study Group
Other: Standard of Care (SOC) — Standard of care
  Arms: Control

SUMMARY:
The goal of this clinical trial is to assess the effect of RenalGuard Therapy in reducing the rates of Acute Kidney Injury (AKI) within 72 hours after cardiac surgery in patients at risk of developing Cardiac Surgery Associated AKI (CSA-AKI) compared to standard-of-care (SoC).

The study is planned to be conducted in 2 clinical sites in the Malaysia - Universiti Malaya Medical Centre and Institut Jantung Negara, Kuala Lumpur, Malaysia.

Participants will be randomized (1:1) to one of the two study groups. The Treatment study group will be managed with the RenalGuard System. The RenalGuard treatment will start after induction of anesthesiology and will run during surgery and for 6-7 hours in the Intensive Care Unit (ICU). The treatment will aim to achieve a urine rate above a predefined urine rate threshold. Patients in the control group will be managed based on the usual clinical practice in cardiac surgery centres as detailed in the recommendations for CSA-AKI prevention by accepted clinical guidelines.

For both study groups general anaesthesia, cardiopulmonary bypass (CPB) run and overall patient care will be based on SoC for cardiac surgery.

Patients will be followed up for up to 7 days post surgery or until discharge, which ever comes first.

Long-term follow up will be performed at 90 days post surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female and >18 years old.
2. Patient able to give written consent.
3. Scheduled for the following non-emergent cardiac surgery procedure requiring CPB, isolated or in combination:

   * coronary artery bypass graft (CABG)
   * aortic valve replacement or repair alone, with or without aortic root repair
   * mitral, tricuspid, or pulmonic valve replacement or repair
   * simultaneous replacement of several cardiac valves
   * CABG with aortic, mitral, tricuspid, or pulmonic valve replacement or repair
   * Surgery on the aorta: aortic root and/ or ascending aorta
   * AF ablation surgery if combined with other cardiac procedures.
   * ASD closure if combined with other cardiac procedures.
   * Excision of myxoma if combined with other cardiac procedures
4. Have at least one of the following risk factors for CSA-AKI:

   * CKD-EPI eGFR 20-59 mL/min/1.73 m²
   * Undergoing combined surgery (e.g. CABG + Valve)
   * STS Score ≥4 or Logistic EuroScore of ≥5 or, Euroscore II of ≥4
   * Left ventricular ejection fraction (LVEF) ≤ 35%
   * Insulin-requiring diabetes
   * Non-insulin-requiring diabetes with HbA1C ≥ 6.1% in the last 6 months
   * Preoperative anemia (hemoglobin ≤11g/dl for men and women) within 4 weeks of surgery

Exclusion Criteria:

1. Patient requiring emergency surgery
2. Surgery to be performed without CPB
3. Patient receiving furosemide at a dose>100 mg/day orally (or the equivalent dose of an alternative loop diuretic) in the last week
4. Patient who cannot be urethrally catheterize for any reason
5. Patients already dialysis dependent
6. Patients with CKD-EPI eGFR <20 mL/min/1.73 m²
7. Known or suspected AKI (KDIGO criteria) at the time of screening
8. IV contrast within 48 hours of surgery
9. Patients participating in another interventional drug or device study or have received an investigational drug or device treatment within the last 30 days
10. Pregnant patient, self-reported
11. Patients whose planned surgery to be performed under conditions of circulatory arrest or hypothermia with rectal temperature < 28°Celsius (82.4° Fahrenheit)
12. Patient with suspected or confirmed bacteraemia, endocarditis, or pyelonephritis at hospital admission
13. Patients with pneumonia, aspiration, or bilateral pulmonary infiltrates from an infectious aetiology reported on chest x-ray or CT scan in the last 7 days
14. Patients in cardiogenic shock or hemodynamic instability which require inotropes or vasopressors or other mechanical devices (Impella, IABP) within 24 hours prior to surgery
15. Patients on extracorporeal membrane oxygenation (ECMO) or durable ventricular assist device (VAD) at the time of screening, or planned use within 24h prior to surgery
16. Patients currently treated with chemotherapy or radiation therapy that may have an impact on kidney function.
17. Patient underwent prior solid organ transplantation
18. Patients underwent major surgery within the last 3 months
19. Any condition which, in the judgement of the investigator, might increase the risk to the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of cardiac surgery-associated acute kidney injury (CSA-AKI) occurring within 72 hours following surgery in the RenalGuard versus Control group | Within 72 hours
  Rate of CSA-AKI as defined by the KDIGO definition i.e. as when any one of the following three criteria are met:
  1. An increase in serum creatinine (SCr) by ≥0.3 mg/dl (≥26.5 umol/l) within 72 hours compared to the baseline value; OR
  2. An increase in SCr by ≥1.5 times from SCr value at baseline within 72 hours; OR
  3. Use of Renal Replacement Therapy (RRT) within 7 days of surgery or by hospital discharge

SECONDARY OUTCOMES:
AKI severity as defined by KDIGO stage definition, with stage distribution between the study groups at 72 hours post-surgery AKI stage | 72 hours
  The staging of AKI (KDIGO) is based on the following criteria:
  Stage 1 Increase ≥ 26 μmol/L within 72 hrs or Increase 1.5 to 1.9 times from baseline
  Stage 2 Increase 2 to 2.9 x reference creatinine
  Stage 3 Increase ≥3 X reference creatinine or increase 354 μmol/L or need for RRT

CONTACTS AND LOCATIONS:
Overall Officials: Krishnasamy Professor Dr. Sivakumar, Principal Investigator — Universiti Malaya Medical Centre
Locations (2):
- Malaysia (2):
  - Institut Jantung Negara, Kuala Lumpur
  - Universiti Malaya Medical Centre, Kuala Lumpur

IPD SHARING:
Plan to Share IPD: Yes
After completion of the study, information regarding the protocol and statistical analysis plan will be shared on request. Additionally anonymised data will be available upon reasonable request.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Luckraz H, Giri R, Wrigley B, Nagarajan K, Senanayake E, Sharman E, Beare L, Nevill A. Reduction in acute kidney injury post cardiac surgery using balanced forced diuresis: a randomized, controlled trial. Eur J Cardiothorac Surg. 2021 Apr 13;59(3):562-569. doi: 10.1093/ejcts/ezaa395. PMID 33236105
- [Background] Redfors B, Bragadottir G, Sellgren J, Sward K, Ricksten SE. Effects of norepinephrine on renal perfusion, filtration and oxygenation in vasodilatory shock and acute kidney injury. Intensive Care Med. 2011 Jan;37(1):60-7. doi: 10.1007/s00134-010-2057-4. Epub 2010 Oct 15. PMID 20949349
- [Background] Brown JK, Shaw AD, Mythen MG, Guzzi L, Reddy VS, Crisafi C, Engelman DT; PeriOperative Quality Initiative and the Enhanced Recovery After Surgery Cardiac Workgroup. Adult Cardiac Surgery-Associated Acute Kidney Injury: Joint Consensus Report. J Cardiothorac Vasc Anesth. 2023 Sep;37(9):1579-1590. doi: 10.1053/j.jvca.2023.05.032. Epub 2023 May 23. PMID 37355415
- [Background] Luckraz H, Giri R, Wrigley B, Hennessy AM, Nicholas J, Nevill A. The use of the RenalGuard system in cardiac surgery with cardiopulmonary bypass: a first in man prospective, observational, feasibility pilot study. Open Heart. 2017 Oct 10;4(2):e000669. doi: 10.1136/openhrt-2017-000669. eCollection 2017. PMID 29071091
- [Background] Lau D, Pannu N, James MT, Hemmelgarn BR, Kieser TM, Meyer SR, Klarenbach S. Costs and consequences of acute kidney injury after cardiac surgery: A cohort study. J Thorac Cardiovasc Surg. 2021 Sep;162(3):880-887. doi: 10.1016/j.jtcvs.2020.01.101. Epub 2020 Mar 3. PMID 32299694
- [Background] Zarbock A, Kullmar M, Ostermann M, Lucchese G, Baig K, Cennamo A, Rajani R, McCorkell S, Arndt C, Wulf H, Irqsusi M, Monaco F, Di Prima AL, Garcia Alvarez M, Italiano S, Miralles Bagan J, Kunst G, Nair S, L'Acqua C, Hoste E, Vandenberghe W, Honore PM, Kellum JA, Forni LG, Grieshaber P, Massoth C, Weiss R, Gerss J, Wempe C, Meersch M. Prevention of Cardiac Surgery-Associated Acute Kidney Injury by Implementing the KDIGO Guidelines in High-Risk Patients Identified by Biomarkers: The PrevAKI-Multicenter Randomized Controlled Trial. Anesth Analg. 2021 Aug 1;133(2):292-302. doi: 10.1213/ANE.0000000000005458. PMID 33684086
- [Background] Mishra PK, Luckraz H, Nandi J, Nevill A, Giri R, Panayiotou A, Nicholas J. Long-term quality of life postacute kidney injury in cardiac surgery patients. Ann Card Anaesth. 2018 Jan-Mar;21(1):41-45. doi: 10.4103/aca.ACA_104_17. PMID 29336390
- [Background] Hoste EAJ, Kellum JA, Selby NM, Zarbock A, Palevsky PM, Bagshaw SM, Goldstein SL, Cerda J, Chawla LS. Global epidemiology and outcomes of acute kidney injury. Nat Rev Nephrol. 2018 Oct;14(10):607-625. doi: 10.1038/s41581-018-0052-0. PMID 30135570
- See also: Related Info — https://kdigo.org/guidelines/acute-kidney-injury/